CLINICAL TRIAL: NCT05737381
Title: Can a Differentiated Oxygen Setup Improve Embryo Quality and Increase the Number of Usable Embryos After in Vitro Fertilization (IVF)?
Brief Title: Quality of Human Embryos in IVF, Culturing in Differentiated Oxygen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Odense Patient Data Explorative Network (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S-20210143
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Infertility; IVF; Embryo
Keywords: Oxygen; Blastocyst; Time lapse; ROS; Embryology
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Sibling study
Who Masked: Participant
Masking Description: Intervention for embryos will be masked when performing the morphokinetic and ROS analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The oocytes from a patient, retrieving more than 8 oocytes will be divided into 2 sibling groups. The control group and the study group.
  The first part of the collected oocytes, will be included as controls. If an unequal numbers of oocytes are collected, the extra oocyte will be included into the control group.
  Control oocytes are, after fertilization, placed in conventional 5% O2 incubators and cultured herein for 5 days.
- Study group (Experimental): The second part of the collected oocytes, from a patient retrieving more than 8 oocytes, will be included as study group.
  Study oocytes, are after fertilization, placed and cultured in conventional 5% O2 incubators for the first 3 days. At day 3, the embryos are moved to an incubator with 2% O2 tension and cultured until day 5.
  Interventions: Other: Differential oxygen tension

INTERVENTIONS:
Other: Differential oxygen tension — By culturing the embryos in a differential O2 set-up, changing the O2 tension from reduced (5% O2) to ultralow (2% O2) from day 3 to day 5 of embryo development in vitro, we mimic the physiological differential changes in O2 as the embryo migrate from the oviduct to the uterus and develops in vivo.
  Arms: Study group

SUMMARY:
The goal of this clinical trial is to evaluate the importance of differential O2 tension to the developing embryos. As a secondary aim, we investigate the levels of reactive oxygen species (ROS) in spent media from the developing blastocysts.

This is a prospective, interventional multicenter study using sibling embryos.

Woman (age 18-41 and normal weight) undergoing assisted reproductive technology (ART) can be included in the study.

Patients included in the project will follow standard IVF protocol and treatment.

By retrieving ≥ 8 oocytes after pickup and upon prior acceptance by the patient, she/the couple can be included in the study.

According to standard treatment, both groups of oocytes will be placed in an incubator with 5% O2.After 3 days of cultivation, the dishes with the study-embryos will be transferred to an incubator with 2% O2. The control embryos will remain in the conventional 5% O2 incubator.

On the fifth day, the embryos will be evaluated, and the blastocyst with expected greatest implantation potential will be transferred to the patients uterus. Surplus embryos with expected implantation potential will be cryopreserved. After transfer or cryopreservation, the media from the wells with used blastocysts will be collected and stored for ROS analysis.

Value for public Health:

If our hypothesis is confirmed, we will be able to optimize the developmental conditions and decreased ROS levels for the embryo in vitro. From a clinical perspective, this could affect the implantation rate of the blastocyst and thus the success of pregnancies for infertile couples while reducing the number of treatments to obtain a viable pregnancy.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the importance of differential O2 tension to the developing embryos. As a secondary aim, we investigate the levels of reactive oxygen species (ROS) in spent media from the developing blastocysts.

This is a prospective, interventional multicenter study using sibling embryos.

Woman (age 18-41 and normal weight) undergoing assisted reproductive technology (ART), with planned IVF or intracytoplasmic sperm injection (ICSI) cycles can be included in the study.

Patients included in the project will follow standard IVF protocol and treatment including hormonal injections, oocyte pick-up, embryo transfer and blastocyst cryopreservation. No further examinations or deviation from standard treatment is necessary in order to participate in the project.

By retrieving ≥ 8 oocytes after pickup and upon prior acceptance by the patient, she/the couple can be included in the study. The minimum number of 8 oocytes has been determined to ensure an average of two blastocysts. The oocytes, will be divided into 2 groups. The first part of the collected oocytes will be included as controls, whereas the second part of the collected oocytes will be included as study group.

According to standard treatment, both groups of oocytes will be placed in an incubator with 5% O2. From time-lapse videos, observations of fertilization and cleavage after 20 hours ± 1h and 44 hours ± 1h, respectively will be annotated. After 3 days of cultivation (68h± 1h), the dishes with the study-embryos will be transferred to a time-lapse incubator with ultralow O2 tension (2%). The control embryos will remain in the conventional 5% O2 time-lapse incubator.

On the fifth day, the embryos will be evaluated by a trained embryologist, and the blastocyst with expected greatest implantation potential will be transferred to the patients uterus. Surplus embryos with expected implantation potential will be cryopreserved. After transfer or cryopreservation, the media from the wells with used blastocysts will be collected and stored for ROS analysis.

Primary outcome:

a) Improved morphokinetics parameters; decreased time difference from 5-cell (t5) to blastocyst stage (tB) in the embryos cultured in differential O2 tensions.

As secondary outcomes:

1. Decreased ROS-activity in spent media from the developing blastocysts cultivated in differential O2 tensions.
2. Number of transferable/vitrified blastocyst in both study and test groups
3. Verification of clinical pregnancy, using ultrasound scanning around week 7. All pregnancies or miscarriage will be registered for all patients if possible.

Value for public Health:

If our hypothesis is confirmed as expected, we will be able to optimize the developmental conditions i.e. faster developmental rate from t5 to tB and decreased ROS levels for the embryo in vitro. From a clinical perspective, this could affect the implantation rate of the blastocyst and thus the success of pregnancies for infertile couples while reducing the number of treatments to obtain a viable pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing assisted reproductive technology (ART), with planned IVF or intracytoplasmic sperm injection (ICSI) cycles.

Women age 18 - 41 years and BMI 18 - 35 kg/m2 (both inclusive) with ≥ 8 oocytes.

Patients will be included no later than at oocyte pick-up.

Exclusion Criteria:

Patients with sperm from testes biopsy, congenital uterine abnormalities, presence of fibromas or polyps, or suspected hydro salpinges. Oocytes from donors.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 350 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Improved morphokinetics parameters | Analysis of morphokinetic, will be finalised approximately 12 months after last intervention.
  Decreased time difference from 5-cell (t5) to full blastocyst stage (tB) in the embryos cultured in differential O2 tensions. This will be analysed using timelapse systems and specific annotation strategies.

SECONDARY OUTCOMES:
Decreased ROS-activity | Analysis of ROS will be finalised approximately 12 months after interventions have been completed.
  Decreased ROS-activity in spent media from the developing blastocysts cultivated in differential O2 tensions. Developing embryos in this project are cultured in seperat wells, allowing for individual analysis of spent media from each unique embryos. After transfer or freezing of embryos, the media is collected and stored for analysis.
Number of transferable/frozen blastocyst | Number count of transferable/vitrified blastocysts will be finalised approximately 6 months after interventions have been complete
  Number of transferable/frozen blastocyst in both control and study group
Clinical pregnancy (CP) | Data of CP from fresh transfers can be finalised 12 months after last intervention. Data of CP from frozen blastocyst can be finalized either within the project or if not used within the following year, in a followup project.
  Number of Clinical pregnancies in both control and study group

CONTACTS AND LOCATIONS:
Overall Officials: Tilde Eskildsen, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided